CLINICAL TRIAL: NCT02920697
Title: Phase I Dose-escalation Study of Oral Administration of the Selective Bcl2 Inhibitor S 55746 in Patients With Refractory or Relapsed Chronic Lymphocytic Leukaemia and B-Cell Non-Hodgkin Lymphoma
Brief Title: Dose-escalation Study of Oral Administration of S 55746 in Patients With Chronic Lymphocytic Leukaemia and B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-55746-001; 2013-003779-36 (EudraCT Number); ISRCTN04804337 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2016-08-23; First posted 2016-09-30 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lymphocytic Leukaemia (CLL); B-Cell Non-Hodgkin Lymphoma (NHL); Multiple Myeloma (MM)
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B-cell Non-Hodgkin Lymphoma (NHL) and Multiple Myeloma (MM) (Experimental)
  Interventions: Drug: S 55746
- Chronic Lymphocytic Leukaemia (CLL) (Experimental)
  Interventions: Drug: S 55746

INTERVENTIONS:
Drug: S 55746 — S 55746, per os administration, from 50 to 1500 mg, once a day during a 21-day cycle. Participants will receive 21-day cycles of treatment until a discontinuation criterion is met.

SUMMARY:
The purpose of this study is to determine the safety profile and tolerability of S 55746 in patients with CLL, B-Cell NHL and MM, in terms of Dose-Limiting Toxicities (DLTs), Maximum Tolerated Dose (MTD) and determine the Recommended Phase 2 Dose (RP2D) through safety profile (DLT, MTD), PK profile, PD profile and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women or men aged >/=18 years
* Patients with a measurable histologically confirmed Follicular Lymphoma (FL), Mantle Cell Lymphoma (MCL), Diffuse Large B-Cell Lymphoma (DLBCL), Small Lymphocytic Lymphoma (SLL) and Marginal Zone Lymphoma (MZL) (Arm A), or patients with an evaluable immunophenotypically confirmed CLL (Arm B), or patients with a measurable Multiple Myeloma t(11;14) (arm A expansion part) according to International Myeloma Working Group (IMWG) criteria
* Relapsed after or refractory disease to standard treatments, and require treatment in the opinion of the investigator
* Estimated life expectancy > 12 weeks
* World Health Organization (WHO) performance status 0-2
* Adequate bone marrow, renal and hepatic functions
* No evidence or treatment for another malignancy within 2 years prior to study entry. Curatively treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia is allowed

Additional inclusion criteria for food interaction cohort:

* B-cell NHL patients at low risk of tumour lysis syndrome (TLS)
* Recent/concomitant treatment altering gastric pH

Exclusion Criteria:

* Previous treatment with a BH3 mimetic
* Previous therapy for the studied disease within 3 weeks before first intake
* Radioimmunotherapy, radiotherapy within 8 weeks before first intake
* Major surgery within 3 weeks before first day of study drug dosing
* Corticosteroids >= 20 mg prednisone equivalent per day within 7 days before first intake
* Anticoagulant oral drugs, aspirin > 325 mg/day within 7 days prior to first S 55746 intake
* Positive direct antiglobulin test (Coombs test) and haptoglobin below normal value
* Prior allogenic stem cell transplant
* Autologous stem cell transplant within 3 months before first intake
* NHL patients diagnosed with Post-Transplant Lymphoproliferative Disease, Burkitt's lymphoma, Burkitt-like lymphoma, or lymphoblastic lymphoma/leukaemia
* Human immunodeficiency virus (HIV)
* Known acute or chronic hepatitis B or hepatitis C
* Impaired cardiac function
* Medications known to prolong corrected QT (QTc) interval
* History or/ clinically suspicious for cancer- related Central Nervous System disease
* Solitary extramedullary plasmacytoma
* Laboratory Signs of TLS
* Strong or moderate CYP3A4 inhibitors/inducers (treatment, food or drink products)
* Treatment highly metabolized by the CYP3A4 or CYP2D6 and/or substrates with a narrow therapeutic index, multienzyme and/or OATP and/or P-gp substrates or herbal products.
* Known hypersensitivity to rasburicase
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency and other cellular metabolic disorders known to cause haemolytic anaemia
* Patients receiving proton pump inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-03; Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During cycle 1 (21 days)
  The MTD is the highest drug dosage that is unlikely (<25% posterior probability) to cause DLT in more than 33% of the treated patients in the first cycle of S 55746 treatment
Incidence of Adverse Events (AEs) | From first dose until 30 days after the last dose intake
  Characterized by severity and seriousness of AEs, laboratory abnormalities and other safety parameters such as electrocardiogram (ECG) changes

SECONDARY OUTCOMES:
Plasma concentration of S 55746 | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D4, C1D5, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
The pharmacokinetic (PK) profile of S 55746: Area Under the Curve [AUC] | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D4, C1D5, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
The PK profile of S 55746: Maximal Concentration [Cmax] | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D4, C1D5, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
Apoptotic activity from blood samples | At Cycle 1(21 days)
Objective Response Rate (ORR) | Up to study completion (maximum of 3 years)
Clinical Benefit Rate (CBR) | Up to study completion (maximum of 3 years)
Duration of response | Up to study completion (maximum of 3 years)
Progression Free Survival (PFS) | From date of inclusion until the date of progression or date of death, whichever occurs first, assessed up to study completion (maximum of 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Le Gouill, M.D., Ph.D., Principal Investigator — Nantes University Hospital
Locations (18):
- The Alfred Hospital Malignant Haematology & Stem Cell Transplantation Services, Melbourne, Australia
- France (4):
  - Hopital Claude Huriez, Lille
  - CHU de Nantes, Nantes
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Gustave Roussy, Villejuif
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Städtisches Klinikum Schwabing, Munich
  - Universitätsklinikum Ulm, Ulm
- Hungary (2):
  - National Oncology Institute, Budapest
  - CRU Hungary Kft, Miskolc
- Poland (2):
  - Warsaw Institute of Oncology, Warsaw
  - Warsaw Medical University, Warsaw
- Singapore (2):
  - National Cancer Center (NCC), Singapore
  - National University Cancer Institute Singapore, Singapore
- South Korea (2):
  - Severance Hospital, Seoul
  - St. Mary's Hospital, Seoul
- United Kingdom (2):
  - University College London Hospitals, London
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Le Gouill S, Wermke M, Morschhauser F, Lim ST, Salles G, Kloos I, de Burgat V, Becquart M, Paux G, Kraus-Berthier L, Pennaforte S, Stilgenbauer S, Walewski J, Ribrag V. A new BCL-2 Inhibitor (S55746/BCL201) as Monotherapy in Patients with Relapsed or Refractory Non-hodgkin Lymphoma: Preliminary Results of the First-in-human Study. Hematol Oncol. 2017 Jun 07;35(S5):14-17. doi: 10.1002/hon.2437_30
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/